CLINICAL TRIAL: NCT03445377
Title: An Open-label, Single-centre, Randomised, Cross-over Design Feasibility Study to Assess the Efficacy of Real-time Continuous Glucose Monitoring in Comparison With Self-monitoring of Blood Glucose in Young Adults and Adolescents With Type 1 Diabetes
Brief Title: Comparison of Real-tiMe ContInuous gLucosE moNitoriNg With Self-monitorIng of Blood Glucose in Young AduLts With Type 1 diabeteS
Acronym: MILLENNIALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R04778
Record Dates: First submitted 2018-02-08; First posted 2018-02-26 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-centre, randomised, crossover design study, involving a 2-week run-in period with blinded CGM, followed by two 8 weeks study periods during which subjects will monitor daily glucose levels either with real-time CGM or SMBG in random order.
Masking Description: This is an open-label, multi-centre, randomised, crossover design study, involving a 2-week run-in period with blinded CGM, followed by two 8 weeks study periods during which subjects will monitor daily glucose levels either with real-time CGM or SMBG in random order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real-time continuous glucose monitoring (Active Comparator): Subjects will be reviewed and a blood sample will be taken for the measurement of HbA1c. Training on the use of DEXCOM G5 or similar will be provided by the research team. Competency on the use of the system will be evaluated. Participants will be advised to use real-time CGM continuously for the next 8 weeks. At the end of the first intervention, a blood sample for the measurement of HbA1c will be taken. Validated questionnaires evaluating diabetes-related distress, management and user acceptance will be completed.
  Interventions: Device: Real-time continuous glucose monitoring
- Self-monitoring of blood glucose (Placebo Comparator): Subjects will be reviewed and a blood sample will be taken for the measurement of HbA1c. During the Control Period, masked CGM will be applied for one week, during Week 1, 4 and 8. At the end of this, a blood sample for the measurement of HbA1c will be taken. Validated questionnaires evaluating diabetes-related distress, management and user acceptance will be completed.
  Interventions: Device: Self-monitoring of blood glucose

INTERVENTIONS:
Device: Real-time continuous glucose monitoring — Subjects randomised to Real-time continuous glucose monitoring will be given a Dexcom G5 or similar, training on its use, and HbA1c measurements taken at the start and end of the study. They will also be given validated questionnaires to complete.
  Arms: Real-time continuous glucose monitoring
Device: Self-monitoring of blood glucose — Subjects randomised to self monitoring of blood glucose will be given a masked CGM which will be applied for one week, during Week 1, 4 and 8. HbA1c measurements will be taken at the start and end of the study. They will also be given validated questionnaires to complete.
  Arms: Self-monitoring of blood glucose

SUMMARY:
The main objective of this study is to determine whether real-time continuous glucose monitoring (CGM) for 8 weeks is more efficacious compared to self-monitoring of blood glucose (SMBG) in young adults with type 1 diabetes.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, randomised, crossover design study, involving a 2-week run-in period with blinded CGM, followed by two 8 weeks study periods during which subjects will monitor daily glucose levels either with real-time CGM or SMBG in random order. Subjects will wear a blinded CGM for a 3-week period during the Control phase. A total of up to 40 subjects (aiming for 30 completed subjects) aged 16 to 24 years with T1D will be recruited through diabetes clinics and other established methods in participating centres. Subjects who drop out of the study within the first 2 weeks of the first intervention period will be replaced.

Subjects will receive appropriate training in the use of real-time CGM. Subjects will have regular contact with the study team during the study.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM. Secondary outcomes are the HbA1c, time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Measures of subject's responses in terms of daily diabetes management, diabetes distress and diabetes technology use and acceptance will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 - 24 years old (inclusive)
2. Type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
3. HbA1c 7.5 - 14.0% based on analysis from local laboratory or equivalent within 1 months of enrolment
4. Treated with insulin pump or MDI
5. Has a Smart phone compatible with Dexcom G5 or similar
6. Willingness to wear study devices
7. Willing to follow study specific instructions
8. Literate in English

Exclusion Criteria:

1. Non-type 1 diabetes mellitus including those secondary to chronic disease
2. Any other physical or psychological disease likely to interfere with the normal conduct of the study
3. Untreated celiac disease or hypothyroidism
4. Current or planned users of real-time or flash (Libre) glucose monitoring sensors
5. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, Metformin, SGLT2 inhibitors, GLP-1 agonists, non-selective beta-blockers and MAO inhibitors etc.
6. Regular use of acetaminophen
7. Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement
8. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which could potentially be used for localisation of the glucose sensor)
9. Lack of reliable telephone facility for contact
10. Known or suspected allergy against insulin
11. Severe visual impairment
12. Severe hearing impairment
13. Subject not proficient in English

Ages: 16 Years to 297 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Sensor Glucose readings within target range | 8 weeks
  Time spent in the target range of 3.9 to 10mmol/l based on sensor glucose levels, throughout the duration of the study periods based on continuous glucose monitoring (CGM).

SECONDARY OUTCOMES:
Sensor Glucose readings below target range | 8 weeks
  Time spent with glucose levels below 3.9 mmol/L based on sensor glucose levels, throughout the duration of the study periods based on continuous glucose monitoring (CGM).
Sensor Glucose readings above target range | 8 weeks
  Time spent with glucose levels above 10.0 mmol/L based on sensor glucose levels, throughout the duration of the study periods based on continuous glucose monitoring (CGM).
HbA1c at 8 weeks | 8 weeks
  HbA1c at 8 weeks (midway point)
Average variation of glucose levels | 8 weeks
  Average variation of glucose levels
Standard deviation variation of glucose levels | 8 weeks
  Standard deviation variation of glucose levels
Coefficient variation of glucose levels | 8 weeks
  Coefficient variation of glucose levels
The time with sensor glucose levels < 3.5 mmol/l , 3.0 and <2.8 mmol/l | 8 weeks
  The time with sensor glucose levels < 3.5 mmol/l , 3.0 and <2.8 mmol/l
The time with sensor glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l) | 8 weeks
  The time with glucose levels in the significant hyperglycaemia (glucose levels > 16.7 mmol/l)
AUC of glucose below 3.5mmol/l | 8 weeks
  AUC (Area under the Curve) of glucose below 3.5mmol/l
Total daily insulin dose | 8 weeks
  Total, basal and bolus insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Hood Thabit, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester Diabetes Centre, Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data such as primary and secondary outcome data will be made available to researchers working directly on the study only.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available within 1 year at the end of study
Access Criteria: Only individuals granted access will be able to view confidential anonymised data from the study.

REFERENCES:
- [Derived] Thabit H, Prabhu JN, Mubita W, Fullwood C, Azmi S, Urwin A, Doughty I, Leelarathna L. Use of Factory-Calibrated Real-time Continuous Glucose Monitoring Improves Time in Target and HbA1c in a Multiethnic Cohort of Adolescents and Young Adults With Type 1 Diabetes: The MILLENNIALS Study. Diabetes Care. 2020 Oct;43(10):2537-2543. doi: 10.2337/dc20-0736. Epub 2020 Jul 28. PMID 32723843